CLINICAL TRIAL: NCT03548129
Title: Empirical Use of Fosfomycin as a Single Dose Oral Treatment of Asymptomatic Bacteriuria
Brief Title: the Use of Fosfomycin as a Single Dose Oral Treatment of Asymptomatic Bacteriuria
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mohammed mahmoud samy, Lecturer in Obstetrics and Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: phosphomycin
Record Dates: First submitted 2016-06-09; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Fosfomycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fosfomycin group (FG) (Active Comparator): Pre-treatment Urine culture will be done then all patients will receive empirical 3 gm oral phosphomycin fosfomycin will be taken by mouth on an empty stomach i.e. 2-3 hours after meals preferably in the evening before bed time after emptying the bladder.
  The contents of 1 packet of Monuril will be dissolved in a glass of water or another non-alcoholic drink and drink immediately. Do not mix with hot water. Do not take fosfomycin in its dry form.
  Response to treatment will be assessed by post-treatment urine culture.
  Interventions: Drug: phosphomycin; Diagnostic Test: Pre-treatment Urine Culture; Diagnostic Test: Post-treatment urine culture
- Culture specific group (CG): (Active Comparator): Pre-treatment Urine culture and antimicrobial sensitivity testing will be done then all patients will receive oral culture specific antibiotic therapy in the form of five days regimen.
  Response to treatment will be assessed by post-treatment urine culture.
  Interventions: Drug: Culture specific antibiotic therapy; Diagnostic Test: Pre-treatment Urine Culture; Diagnostic Test: Antimicrobial sensitivity testing; Diagnostic Test: Post-treatment urine culture

INTERVENTIONS:
Drug: phosphomycin — Single dose 3 gm oral fosfomycin will be taken by mouth on an empty stomach
  Arms: Fosfomycin group (FG)
Drug: Culture specific antibiotic therapy — Culture-specific antibiotic treatment for 5 days
  Arms: Culture specific group (CG):
Diagnostic Test: Pre-treatment Urine Culture — Mid-stream urine sample will be cultured and number of CFU per mL will be determined.
Diagnostic Test: Antimicrobial sensitivity testing — Susceptibility of urinary pathogens to various antimicrobials
  Arms: Culture specific group (CG):
Diagnostic Test: Post-treatment urine culture — Mid-stream urine sample will be cultured and number of CFU per mL will be determined.

SUMMARY:
Urinary tract infections (UTIs) are the most commonly occurring bacterial infections in women, Asymptomatic bacteriuria (AB) is a common complication during pregnancy, with a prevalence of 2-10%. It has been associated with a greater incidence of symptomatic urinary tract infection (UTI), as well as foetal and obstetric complications. Appropriate treatment reduces the incidence of UTI by 80-90%, as well as the risk of a premature birth and low-birth-weight baby Fosfomycin trometamol (Monuril) is approved in numerous countries worldwide, including various European countries and the USA, mainly for the treatment of uncomplicated UTIs

DETAILED DESCRIPTION:
This study aims to compare between the efficacy of empirical use of fosfomycin trometamol and the use of selected antimicrobials according to urinary culture and sensitivity in curing asymptomatic bacteriuria.

All women included in the study will be counseled regarding mode of intervention and informed consent will be obtained. All cases will be subjected to complete history taking, routine antenatal examination and investigations including complete blood picture, kidney functions and urine analysis, treatment of genital infection if diagnosed. Routine obstetric ultrasound examination.

Patients will be randomized into two groups:

1. Group (A): Fosfomycin group (FG); where all patients will receive empirical 3 gm oral fosfomycin fosfomycin will be taken by mouth on an empty stomach i.e. 2-3 hours after meals preferably in the evening before bed time after emptying the bladder.

   The contents of 1 packet of Monuril will be dissolved in a glass of water or another non-alcoholic drink and drink immediately. Do not mix with hot water. Do not take fosfomycin in its dry form.

   Nature: also known as phosphomycin, phosphonomycin, is a broad-spectrum antibiotic, produced by certain Streptomyces species, although it can now be made by chemical synthesis.

   Trade name: Monuril Company: Zambon, Pharma Con Company, Switzerland
2. Group (B): Culture specific group (CG): where all patients will receive oral antibiotic according to urine culture and sensitivity, oral antibiotics will be given in the form of five days regimen.

How the urine sample will be collected? The caregiver will give the patient a sterile cup and lid, and advice her to wash herself completely then clean the perineal area from anterior to posterior by water and in standing position as male begin to urinate then stop urinating put the sterile cup and catch the rest of urine in it. Do not touch the inside of the cup or the lid. Put the lid on the cup.

One week after completing the course of treatment all patients included in the study will be subjected to colony count evaluation, to figure out the need for:

1. Urine culture in fosfomycin group in case of inadequate response to treatment and to give antibiotic according.
2. The change of duration or the type of antibiotic in case of inadequate response to initial treatment in the culture group.

Outcomes

Primary:

* Resolution of asymptomatic bacteriuria as measured by colony count.
* Time frame: 1 week

Secondary:

1. Side effects of fosfomycin as, nausea, diarrhea, headache, vaginal itching, runny nose, back pain Side effects from other antibiotics in culture and sensitivity group
2. Need for further treatment, either extending the course of treatment into 5 or 7 days regimen or changing the antibiotic in case of inadequate initial response.
3. Need for further investigations, as urine culture and sensitivity for fosfomycin group in case of inadequate response on empirical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant patients from 13 weeks to 36 weeks gestation.
2. Pus cells in urine analysis >5/HPF.
3. ≥ 105 colony-forming units (CFU) per millilitre of the same microorganisms in two consecutive cultures.
4. No symptoms or sings suggestive of urinary tract infection.

Exclusion Criteria:

1. Presence of any urinary symptoms as burning micturition, hesitancy
2. Fever and loin pain.
3. Diabetes mellitus.
4. Known to be allergic from any of the antimicrobial ingredients.
5. Not using any antimicrobial during the course of treatment for any other infection.
6. Not known to have any congenital urinary anomalies.
7. If the patient is taking medications that interact with fosfomycin as:

   * Anorexiants (eg, phentermine) or certain sympathomimetics (eg, albuterol, amphetamine, pseudoephedrine) because the risk of their side effects may be increased by fosfomycin.
   * Lithium or tetracyclines because their effectiveness may be decreased by fosfomycin.
   * Metoclopramide because it may decrease fosfomycin's effectiveness.
8. Impaired kidney functions (creatinine's clearance is <80 ml/min.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Resolution of asymptomatic bacteriuria | 1 week
  Decline in colony forming unit (CFU)/mL or absence of bacterial growth after treatment

SECONDARY OUTCOMES:
Need for further treatment | 1 week
  Either extending the course of treatment into 5 or 7 days regimen or changing the antibiotic in case of inadequate initial response.
Need for further investigations | 1 week
  Need for urine culture and sensitivity in fosfomycin group in case of inadequate response on empirical treatment.
Incidence of adverse drug reactions . | 1 week
  Incidence of adverse drug reactions as nausea, diarrhea, headache, vaginal itching, runny nose, back pain Side effects from other antibiotics in culture and sensitivity group

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Samy, MD, Principal Investigator — M Samy

IPD SHARING:
Plan to Share IPD: No